CLINICAL TRIAL: NCT03423875
Title: Predicting Emergency Department Delirium With an Interactive Customizable Tablet to Prevent Repeat Visits (PrEDDICT-PReV) App
Brief Title: Predicting Emergency Department Delirium With an Interactive Customizable Tablet to Prevent Repeat Visits
Acronym: PrEDDICT-PReV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 269-2017
Record Dates: First submitted 2017-12-20; First posted 2018-02-06 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Delirium
Keywords: Delirium, Delirium Recognition
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: To prevent outcome assessment bias, research staff will be masked as to the randomization status of participants until after they have completed and recorded gold-standard delirium assessments of delirium using the Confusion Assessment Method .
  Similarly, ED physicians will be blinded to the gold standard assessments of delirium made by research assistants as well as the results of the PrEDICT test scores when they make their baseline clinical assessments of delirium. ED Physicians will also remain masked until they have recorded their discharge plan. The intervention focuses on the impact of revealing the result of the PrEDICT game scores on ED physicians' recognition of delirium, so randomization status must be revealed to them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients assigned to the control condition will be treated using the current standard of care, clinical assessments, to identify delirium.
- Intervention (Experimental): PrEDICTgame score (subject's relative risk of delirium) will be shared with ED physicians in the intervention arm. After viewing the tests results, ED physicians will be asked to reassess delirium risk, and indicate if they would change their management based on the PrEDICT app scores.
  Interventions: Diagnostic Test: PrEDICT game score

INTERVENTIONS:
Diagnostic Test: PrEDICT game score — PrEDICT game score will be shared with the emergency physicians and health care professionals
  Arms: Intervention

SUMMARY:
Delirium is a common and serious complication of medical care that affects 10% of older Emergency Department (ED) patients, which unfortunately is unrecognized in up to 75% of ED patients.Studies have shown that 26 - 42% of patient with delirium are sent home. And 80% of patients sent home with unrecognized delirium are re-hospitalized within 4 days. Unrecognized delirium also has grave consequences for patient care - Kakuma showed that patient with unrecognized delirium who were sent home had 3-8x the mortality rate of patients with recognized delirium at 6 months.

Fluctuating severity over time is a key clinical characteristics of delirium, making its diagnosis challenging. Regardless of cause, failure to recognize delirium means that ED staff cannot meet their patient"s needs. For example, ED staff may miss serious medical conditions associated with delirium, may not provide understandable discharge instructions or ensure a caregiver can supervise and assist a patient with delirium who is discharged. These care adaptations require staff to recognize the presence of delirium. Thus it is not surprising that unrecognized delirium has such grave consequences for patients.

Thus recognition of delirium is critical to improving patient outcomes and reducing repeat ED visits. Patients with delirium may appear to have normal mental status at times, making its diagnosis challenging. High levels of service demand in the ED, plus the competing demands of numerous other initiatives to improve quality and reduce waiting times may explain why delirium continue to go unrecognized despite guidelines promoting routine delirium screening as a top priority in the ED. To address this care gap, the investigators developed an innovative solution. Rather than adding tasks to overburdened ED staff, our solution takes advantage of the long waiting times clients have in the ED for their initial assessments and between interactions with clinical staff. During these times, patients will use the PrEDICT "serious game" - similar to the Whack-a-Mole carnival game. The investigators have developed an algorithm based on participants" performance on this simple but serious game that can identify patients at high risk for delirium.

The investigators propose to conduct a prospective, multi-center randomized clinical trial in 4 provinces. The primary objective of this study is to assess the impact of our tablet technology on the recognition of delirium by ED staff. All eligible patients who agree to participate will be treated in the same manner and will play the PrEDICT tablet based game. The investigators will randomly assign half of patients to have their test performance shared with clinical staff. Patients assigned to the control condition will be treated using the current standard of care, clinical assessments, to identify delirium.

This project will allow us to solidly advance this technology from a working prototype (TRL7) to a commercially ready product demonstrated effective in multiple "real-world" environments under expected operational conditions (TRL8). Also it will provide evidence that the PrEDICT tablet app is clinically, technically, commercially and operationally feasible.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age and older
* Have been in the ED for a minimum of 4 hours at the time of screening

Exclusion Criteria:

* Live in a full care nursing home
* Have a critical illness (Canadian Triage Acuity Score rendering them unable to communicate or provide consent)
* Have delirium prior to ED arrival
* Do not assent to study participation
* Have visual impairment that makes them unable to use the serious game tablet
* Have other communication difficulties preventing use of the serious game tablet

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1375 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Delirium recognition by ED staff | Delirium recognition by ED staff will be measured during their index ED visit, within 4 hours of assessment using the PrEDICT app.
  Design a simple dichotomous question to assess whether MD's clinically diagnose the presence of delirium in a specific patient(not delirious vs. delirious). In addition, ask MD's to rate their certainty of their diagnosis on a 10 point Numeric Rating scale. The primary outcome will be determined based on the dichotomous question

SECONDARY OUTCOMES:
Ability of the PrEDICT app to identify patients with incident delirium | Between 7-14 days of ED discharge
  Our Secondary outcome will be to correlate the PrEDICT game score with patients who develop incident delirium as assessed using the CAM
Ability of the PrEDICT app to identify patients at high risk for incident delirium | Between 7-14 days of ED discharge
  Our Secondary outcome will be to correlate the PrEDICT game score with patients who develop incident delirium as assessed using delirium index
Unanticipated Barriers to using the PrEDICT app | Day 1(ED visit) to Day 4
  Clinical feasibility will be assessed as the proportion of eligible patients that are able to complete use of the PrEDICT serious game.
Feasibility of Tablet Administration by Other Stakeholders | Day 1(ED visit) to Day 4
  In patients who have already completed the main study and primary outcome, a convenience subsample will be recruited to compare the relative completion rate of the PrEDICT app by patients who are being supervised by: i) nurses; ii) trained hospital volunteers; and iii) family members and care givers.

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - Nova Scotia Health Authority, Nova Scotia, Halifax
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - CHU de Québec - Université Laval, Québec, Quebec
  - Alberta Health Services, Calgary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hustey FM, Meldon SW. The prevalence and documentation of impaired mental status in elderly emergency department patients. Ann Emerg Med. 2002 Mar;39(3):248-53. doi: 10.1067/mem.2002.122057. PMID 11867976
- [Background] Kakuma R, du Fort GG, Arsenault L, Perrault A, Platt RW, Monette J, Moride Y, Wolfson C. Delirium in older emergency department patients discharged home: effect on survival. J Am Geriatr Soc. 2003 Apr;51(4):443-50. doi: 10.1046/j.1532-5415.2003.51151.x. PMID 12657062
- [Background] Adamis D, Treloar A, Darwiche FZ, Gregson N, Macdonald AJ, Martin FC. Associations of delirium with in-hospital and in 6-months mortality in elderly medical inpatients. Age Ageing. 2007 Nov;36(6):644-9. doi: 10.1093/ageing/afm094. Epub 2007 Jul 28. PMID 17660528
- [Background] McCusker J, Cole M, Abrahamowicz M, Primeau F, Belzile E. Delirium predicts 12-month mortality. Arch Intern Med. 2002 Feb 25;162(4):457-63. doi: 10.1001/archinte.162.4.457. PMID 11863480
- [Background] Lewis LM, Miller DK, Morley JE, Nork MJ, Lasater LC. Unrecognized delirium in ED geriatric patients. Am J Emerg Med. 1995 Mar;13(2):142-5. doi: 10.1016/0735-6757(95)90080-2. PMID 7893295
- [Background] Elie M, Rousseau F, Cole M, Primeau F, McCusker J, Bellavance F. Prevalence and detection of delirium in elderly emergency department patients. CMAJ. 2000 Oct 17;163(8):977-81. PMID 11068569
- [Background] Hustey FM, Meldon S, Palmer R. Prevalence and documentation of impaired mental status in elderly emergency department patients. Acad Emerg Med. 2000 Oct;7(10):1166. PMID 11015259
- [Background] Monette J, Galbaud du Fort G, Fung SH, Massoud F, Moride Y, Arsenault L, Afilalo M. Evaluation of the Confusion Assessment Method (CAM) as a screening tool for delirium in the emergency room. Gen Hosp Psychiatry. 2001 Jan-Feb;23(1):20-5. doi: 10.1016/s0163-8343(00)00116-x. PMID 11226553
- [Background] Schuurmans MJ, Duursma SA, Shortridge-Baggett LM. Early recognition of delirium: review of the literature. J Clin Nurs. 2001 Nov;10(6):721-9. doi: 10.1046/j.1365-2702.2001.00548.x. PMID 11822843
- [Background] Hustey FM, Meldon SW, Smith MD, Lex CK. The effect of mental status screening on the care of elderly emergency department patients. Ann Emerg Med. 2003 May;41(5):678-84. doi: 10.1067/mem.2003.152. PMID 12712035
- [Background] Wilber ST, Carpenter CR, Hustey FM. The Six-Item Screener to detect cognitive impairment in older emergency department patients. Acad Emerg Med. 2008 Jul;15(7):613-6. doi: 10.1111/j.1553-2712.2008.00158.x. PMID 18691212
- [Background] Han JH, Zimmerman EE, Cutler N, Schnelle J, Morandi A, Dittus RS, Storrow AB, Ely EW. Delirium in older emergency department patients: recognition, risk factors, and psychomotor subtypes. Acad Emerg Med. 2009 Mar;16(3):193-200. doi: 10.1111/j.1553-2712.2008.00339.x. Epub 2009 Jan 20. PMID 19154565
- [Background] Carpenter CR, Bassett ER, Fischer GM, Shirshekan J, Galvin JE, Morris JC. Four sensitive screening tools to detect cognitive dysfunction in geriatric emergency department patients: brief Alzheimer's Screen, Short Blessed Test, Ottawa 3DY, and the caregiver-completed AD8. Acad Emerg Med. 2011 Apr;18(4):374-84. doi: 10.1111/j.1553-2712.2011.01040.x. PMID 21496140
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] McCusker J, Cole MG, Dendukuri N, Belzile E. The delirium index, a measure of the severity of delirium: new findings on reliability, validity, and responsiveness. J Am Geriatr Soc. 2004 Oct;52(10):1744-9. doi: 10.1111/j.1532-5415.2004.52471.x. PMID 15450055
- [Background] Sylvestre MP, McCusker J, Cole M, Regeasse A, Belzile E, Abrahamowicz M. Classification of patterns of delirium severity scores over time in an elderly population. Int Psychogeriatr. 2006 Dec;18(4):667-80. doi: 10.1017/S1041610206003334. Epub 2006 Apr 27. PMID 16640798
- [Background] Zou Y, Cole MG, Primeau FJ, McCusker J, Bellavance F, Laplante J. Detection and diagnosis of delirium in the elderly: psychiatrist diagnosis, confusion assessment method, or consensus diagnosis? Int Psychogeriatr. 1998 Sep;10(3):303-8. doi: 10.1017/s1041610298005390. PMID 9785149